CLINICAL TRIAL: NCT03272451
Title: ECG-guided Immediate pRimAry Percutaneous Coronary Intervention for Culprit Vessel Using a Transradial Single Guiding Catheter to Reduce Door to Device Time: RAPID II Study
Brief Title: ECG-guided Immediate Primary PCI for Culprit Vessel to Reduce Door to Device Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Luhe Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BeijingLH
Record Dates: First submitted 2017-08-30; First posted 2017-09-05 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- culprit vessel intervention (Experimental): culprit vessel PCI prior to contralateral angiography using a single transradial guiding catheter
  Interventions: Procedure: culprit vessel intervention
- traditional approach (Active Comparator): complete coronary angiography followed by guiding catheter selection for culprit vessel PCI
  Interventions: Procedure: traditional approach

INTERVENTIONS:
Procedure: culprit vessel intervention — ECG guided immediate culprit vessel intervention using a single transradial guiding catheter such as MAC or JL 3.5
  Arms: culprit vessel intervention
Procedure: traditional approach — single diagnostic catheter for complete coronary angiography and guiding catheter selection for PCI
  Arms: traditional approach

SUMMARY:
No consensus exists about which coronary artery should be firstly catheterized in primary percutaneous coronary intervention (PCI). The aim of the present study was to compare door-to-balloon time (D2B) of ECG guided immediate infarct-related artery (IRA) PCI with traditional complete coronary angiography followed by PCI for the treatment of ST segment elevation myocardial infarction (STEMI) patients. Primary endpoint is door to device (D2D) time. Secondary end-points are: puncture to device (P2D) time,first medical contact to device (FMC2D) time,incidence of radial artery spasm and occlusion, contrast amount, fluoroscopy time, cumulative air kerma(CAK) and dose area product(DAP).

ELIGIBILITY:
Inclusion Criteria:

* Patient must be > 18 years of age
* Patients have typical chest pain for at least 20 minutes and have ECG changes typical for STEMI (ST elevation≥2mm in two continuous precordial leads or ST elevations≥1mm in two limb leads or new left bundle branch block) or ECG changes compatible with true posterior MI
* Symptoms ≥ 30 min and ≤12 hours
* Patient and treating interventional cardiologist agree for randomization
* Patient provides written informed consent
* Diagnostic and therapeutic intervention performed through transradial artery approach
* Palpable radial artery.

Exclusion Criteria:

* Concurrent participation in other investigational study
* Current platelet count <100 x 10^9cells/L or Hgb <10 g/dL
* Absence of radial artery pulsation
* Active bleeding or significant increased risk of bleeding, severe hepatic insufficiency, current peptic ulceration, proliferative diabetic retinopathy
* Uncontrolled hypertension
* Prior CABG surgery
* Fibrinolytic therapy for current MI treatment
* patient have a life expectancy of <180days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
door to device (D2D) time | 24hours
  time patient's arrival at our hospital to first device (balloon,aspiration catheter or stent) use

SECONDARY OUTCOMES:
puncture to device (P2D) time | 24hours
  time from radail artery puncture to first device(balloon,aspiration catheter or stent) use
first medical contact to device (FMC2D) time | 24hours
  time from first medical contact to first device (balloon,aspiration catheter or stent) use.
incidence of radial artery spasm | during the procedure (time from the guide catheter inserted to guide catheter removed)
  radial artery spasms were defined as follows. Severe, moderate, and mild based on radiao angiography before and after procedure
incidence of radial artery occlusion | inhospital (an expected average of 5 days),30day,12month
  the absence of palpable radial artery pulsation confirmed by echocardiogram
fluoroscopy time | 1 hour
  recorded on the machine
cumulative air kerma(CAK) and dose area product(DAP). | 1 hour
  recorded on the machine

OTHER OUTCOMES:
MACE | 12 month
  major advance cardiac event (MACE)including cardiacdeath, myocardial infarction (MI) and target vessel revascularization (TVR)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Luhe hospital, Beijing, China

REFERENCES:
- [Derived] Guo J, Wang G, Li Z, Liu Z, Wang Y, Wang S, Wang Y, Wu Y, Wang H, Wang Y, Zhang L, Hua Q. Culprit vessel revascularization first with primary use of a dedicated transradial guiding catheter to reduce door to balloon time in primary percutaneous coronary intervention. Front Cardiovasc Med. 2022 Oct 28;9:1022488. doi: 10.3389/fcvm.2022.1022488. eCollection 2022. PMID 36386357